CLINICAL TRIAL: NCT01085682
Title: Application and Effectiveness Analysis of Internet-based Diabetes Prevention Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kun-Ho Yoon, Professor, Medical doctor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KCMC07OT255
Record Dates: First submitted 2010-02-19; First posted 2010-03-12 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes prevention; Lifestyle modification; Obesity; Impaired glucose tolerance; Diet; Physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Glucose Intolerance; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Lifestyle counseling
- Standard care (Active Comparator)
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Lifestyle counseling — In intervention group, counseling sessions are conducted weekly for 3 months, once per two weeks for 3 months, monthly for 18 months, and then once every two months for the remainder of the study.
  Arms: Lifestyle counseling
Behavioral: Standard care — In standard care group, counseling sessions are conducted only 6 times for 4 years
  Arms: Standard care

SUMMARY:
This study was conducted to test the possibility of preventing or delaying the development of type 2 diabetes in individuals with impaired glucose tolerance and elevated fasting plasma glucose concentrations by internet-based diabetes prevention program.

DETAILED DESCRIPTION:
Diabetes is common and rapidly increasing, because of obesity, unhealthy eating habits, and physical inactivity in Korea. Many studies reported that lifestyle modification related in the primary prevention of diabetes in multiethnic populations. The aim of this study is to determine whether internet-based interventions in those at high risk may delay the development of type 2 diabetes mellitus, and thereby reduce the incidence of cardiovascular diseases and strokes in Korean populations. In January 2008, participant recruitment began in Chung-ju city, a rural area in Korea. The subjects with impaired glucose tolerance or elevated fasting plasma glucose concentrations were selected from initial screening and then randomized to either a control or intensive lifestyle group to carry out intervention over 4 years. The primary outcome of this study is the development of diabetes by ADA criteria. To confirm the onset of diabetes, all subjects have an OGTT at the interim 6-month and each annual visit. Also, systematic evaluation examination will be done at the same time. The proportion of subjects developing diabetes in each group and the factors relating the progression will be estimated using statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age of 30-69 years
* BMI ≥ 20 kg/m2
* Impaired glucose tolerance :

  2h postprandial glucose (75 g OGTT) 140-199 mg/dl or Impaired fasting glucose : Fasting plasma glucose 110-125 mg/dl

Exclusion Criteria:

* Diabetes at baseline
* Cardiovascular disease, cancer requiring treatment in the past 5 years, renal disease
* Unable to communicate with clinic staff, Pregnancy and childbearing

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, M.D., Ph.D., Study Director — Kangnam St.Mary's hospital
Locations (1):
- Chung-ju health care center, Chungju, Chungchungbook-do, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Counseling | Standard Care
Started | 31 | 28
Completed | 6 | 3
Not Completed | 25 | 25
Not completed — Withdrawal by Subject | 25 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Standard Care | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (3) | 55 (3) | 55 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Type 2 Diabetes Mellitus
Description: Incidence of type 2 diabetes mellitus
Time Frame: one year follow up
Measure: Number; unit: participants
Arm/Group | Lifestyle Counseling | Standard Care
Number analyzed (Participants) | 6 | 3
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Lifestyle Counseling | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No